CLINICAL TRIAL: NCT03552939
Title: The Power of Maternal Microbes on Infant Health
Brief Title: The Impact of Maternal Microbes on Infant Health Programming
Acronym: MAMI
Status: Completed | Type: Observational
Sponsor: Institute of Agrochemistry and Food Technology, National Research Council (Other Government)
Collaborators: Fundación para la Investigación del Hospital Clínico de Valencia (Other); Hospital Universitario La Fe (Other); Hospital de Manises (Other); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other); CS Serreria II (Unknown); CS La Eliana (Unknown)
Responsible Party: Principal Investigator, Maria Carmen Collado, Principal Investigator, Institute of Agrochemistry and Food Technology, National Research Council
Other Study IDs: 639226
Record Dates: First submitted 2018-03-21; First posted 2018-06-12 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: microbiota; breast milk; diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
MAMI aims to characterize maternal microbes to be transferred to neonates and determine their function in infant health programming.

DETAILED DESCRIPTION:
Recent reports suggest that early microbial colonization has an important role for in promoting health. This may contribute to reduce the risk of chronic diseases such as obesity, allergies and inflammatory conditions. Advances in understanding host-microbe interactions imply that maternal microbiota plays a crucial role on health programming. This process begins in utero and it is modulated by mode of delivery and diet. The investigator's previous data has shown that i) specific shifts in milk microbial composition are associated with lactation time and mode of delivery, ii) milk microbes drive the infant microbiota composition; iii) maternal microbiota dysbiosis may be transferred to the infant. However, factors defining maternal microbiota and its biological role upon infant's health are not yet fully understood. Hence, this project aims to characterize maternal microbes to be transferred to neonates and determine their function in infant health programming. The specific aims are:(1) understanding how the maternal microbiome is influenced by host and environmental factors;(2) characterizing the microbial core and bioactive compounds transmitted to the offspring mainly via breastfeeding and their key roles in the microbial modulation and host response;(3) understanding the interactions among breast milk bioactive compounds and their role in infant health;(4) shedding light on how maternal microbes influence the infant immune system.

Results obtained will demonstrate the interaction between infant nutrition, microbes and host response in early life and its key role in health programming, enabling new applications in the field of personalized nutrition & medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* Healthy woman (no medication, no diabetes, no pre-gestational thyroid problems)
* Postpartum woman (beginning of the puerperium).

Exclusion criteria:

* Non-compliance with any of the inclusion criteria.
* Medication and drugs
* Health problems at the immunological and metabolic levels.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women (pregnant women)
Study Population: Families located on the Mediterranean area
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Microbiota composition | from birth to 24 month
  Dominant microbial species maternal and infant samples (using qPCR and sequencing -approaches analysis

SECONDARY OUTCOMES:
Maternal diet | from birth to12 month
  Maternal diet (FFQ) during gestation and 12 month post-partum
Maternal BMI | pre-gestational
  To check Body Mass Index (kg/cm2)
Maternal weight | pre-gestational and from birth to 12 months post-partum
  To check Weight gain over pregnancy (kg) and weight during lactation
To identify maternal factors affecting microbiota: antibiotics | pre-gestational
  antibiotics treatment during gestation (number of treatments)
To identify the impact of mode of delivery | Birth
  Mode of delivery type: Vaginal/C-section (elective or non-elective)
Infant weight | from birth to 24 month
  Infant weight (kg)
Infant height | from birth to 24 month
  Infant height (cm)
Infant Diet | from bith to 24 month
  Exclusive breastfeeding time (months), breastfeeding duration and time of introduction of complementary food
Fecal short-chain fatty acids | from birth to 24 month
  Determine the relationship between fecal microbiota composition and fecal short chain fatty acids

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Fundacion Investigacion Sanitaria INCLIVA, Valencia
  - Hospital Universitario y Politecnico la Fe, Valencia

REFERENCES:
- [Result] Boix-Amoros A, Martinez-Costa C, Querol A, Collado MC, Mira A. Multiple Approaches Detect the Presence of Fungi in Human Breastmilk Samples from Healthy Mothers. Sci Rep. 2017 Oct 12;7(1):13016. doi: 10.1038/s41598-017-13270-x. PMID 29026146
- [Result] Gomez-Gallego C, Kumar H, Garcia-Mantrana I, du Toit E, Suomela JP, Linderborg KM, Zhang Y, Isolauri E, Yang B, Salminen S, Collado MC. Breast Milk Polyamines and Microbiota Interactions: Impact of Mode of Delivery and Geographical Location. Ann Nutr Metab. 2017;70(3):184-190. doi: 10.1159/000457134. Epub 2017 Mar 17. PMID 28301837
- [Result] Kumar H, du Toit E, Kulkarni A, Aakko J, Linderborg KM, Zhang Y, Nicol MP, Isolauri E, Yang B, Collado MC, Salminen S. Distinct Patterns in Human Milk Microbiota and Fatty Acid Profiles Across Specific Geographic Locations. Front Microbiol. 2016 Oct 13;7:1619. doi: 10.3389/fmicb.2016.01619. eCollection 2016. PMID 27790209
- [Result] Boix-Amoros A, Collado MC, Mira A. Relationship between Milk Microbiota, Bacterial Load, Macronutrients, and Human Cells during Lactation. Front Microbiol. 2016 Apr 20;7:492. doi: 10.3389/fmicb.2016.00492. eCollection 2016. PMID 27148183
- [Derived] Flores Ventura E, Bernabeu M, Callejon-Leblic B, Cabrera-Rubio R, Yeruva L, Estan-Capell J, Martinez-Costa C, Garcia-Barrera T, Collado MC. Human milk metals and metalloids shape infant microbiota. Food Funct. 2024 Dec 9;15(24):12134-12145. doi: 10.1039/d4fo01929f. PMID 39584920
- [Derived] Yeruva L, Mulakala BK, Rajasundaram D, Gonzalez S, Cabrera-Rubio R, Martinez-Costa C, Collado MC. Human milk miRNAs associate to maternal dietary nutrients, milk microbiota, infant gut microbiota and growth. Clin Nutr. 2023 Dec;42(12):2528-2539. doi: 10.1016/j.clnu.2023.10.011. Epub 2023 Oct 16. PMID 37931372
- [Derived] Selma-Royo M, Calatayud Arroyo M, Garcia-Mantrana I, Parra-Llorca A, Escuriet R, Martinez-Costa C, Collado MC. Perinatal environment shapes microbiota colonization and infant growth: impact on host response and intestinal function. Microbiome. 2020 Nov 23;8(1):167. doi: 10.1186/s40168-020-00940-8. PMID 33228771
- [Derived] Cortes-Macias E, Selma-Royo M, Garcia-Mantrana I, Calatayud M, Gonzalez S, Martinez-Costa C, Collado MC. Maternal Diet Shapes the Breast Milk Microbiota Composition and Diversity: Impact of Mode of Delivery and Antibiotic Exposure. J Nutr. 2021 Feb 1;151(2):330-340. doi: 10.1093/jn/nxaa310. PMID 33188413
- [Derived] Selma-Royo M, Garcia-Mantrana I, Calatayud M, Parra-Llorca A, Martinez-Costa C, Collado MC. Maternal diet during pregnancy and intestinal markers are associated with early gut microbiota. Eur J Nutr. 2021 Apr;60(3):1429-1442. doi: 10.1007/s00394-020-02337-7. Epub 2020 Jul 29. PMID 32728880
- [Derived] Garcia-Mantrana I, Alcantara C, Selma-Royo M, Boix-Amoros A, Dzidic M, Gimeno-Alcaniz J, Ubeda-Sansano I, Sorribes-Monrabal I, Escuriet R, Gil-Raga F, Parra-Llorca A, Martinez-Costa C, Collado MC; MAMI team. MAMI: a birth cohort focused on maternal-infant microbiota during early life. BMC Pediatr. 2019 May 3;19(1):140. doi: 10.1186/s12887-019-1502-y. PMID 31053102